CLINICAL TRIAL: NCT05578898
Title: CLEAR Care Companion Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2021.077; HUM00201652 (Other: University of Michigan)
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer; Radical Cystectomy
Keywords: Mobile application; Post surgical care
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLEAR CC (Experimental): Patients use CLEAR CC application with Smartphone or Tablet
  Interventions: Behavioral: CLEAR Care Companion (CC) application

INTERVENTIONS:
Behavioral: CLEAR Care Companion (CC) application — The CLEAR CC application is an EPIC-based, electronic application, downloaded to the patient's Smartphone or Tablet. The CLEAR CC leverages patient-reported symptoms assessment vis-a-vis push notifications to complete clinically meaningful questions and validated questionnaires pertaining to symptoms that serve as early indicators of readmission. The CLEAR CC application will send notifications beginning two days prior to surgery and continue until the 6 week post operative appointment.

SUMMARY:
Hospital readmissions are common after major cancer surgery, leading to poorer patient outcomes, increased mortality and additional costs. In this study, Clinical and Engineering Approaches to Readmission (CLEAR) Care Companion Application, investigators aim to utilize a smartphone application that tracks concerning postoperative symptoms and provides educational interventions to determine if this can minimize delays in communication between patients and medical providers, increase patient satisfaction with the care received, and reduce or lessen the severity of readmissions.

DETAILED DESCRIPTION:
Patients complete clinically meaningful questions and validated questionnaires pertaining to physiological and psychological symptoms that serve as early indicators of readmission, with the aim to improve experience by empowering patient to be active participants in their recovery, identify complications early to minimize morbidity and reduce overall readmissions.

The study has the following three objectives: (1) Assess patient engagement with the CLEAR Care Companion application for patients that have undergone radical cystectomy (2) Measure patient experience with the application and its effect on satisfaction with overall care (3) Evaluate the effect of the application on case complexity (readmission intensity) and overall readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a radical cystectomy with reconstruction through GU Oncology Clinic
* Patient at the University of Michigan (Michigan Medicine)
* Access to compatible smartphone or tablet device

Exclusion Criteria:

* Non-English speaking patients
* Patients without access to a smart phone or tablet with internet capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Frequency of engagement with application | 42 days post hospital discharge
  To measure patient engagement with the application, the number of responses to application notifications and patient inputs will be captured in the electronic medical record (EMR). Descriptive statistics will be used to assess frequency and duration of engagement.
Duration of engagement with application | 42 days post hospital discharge
  To measure patient engagement with the application, the number of responses to application notifications and patient inputs will be captured in the electronic medical record (EMR). Descriptive statistics will be used to assess frequency and duration of engagement.
Patient Experience Survey -- Overall Care (all participants) | 42 days post hospital discharge
  Assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS®) GLOBAL 10 questionnaire.
Patient Experience Survey -- Overall Care (first 20 participants) | 42 days post hospital discharge
  The first 20 participants will complete a qualtrix survey.
Readmission intensity | 42 days post hospital discharge
  To measure the change in complexity of readmissions (readmission intensity), readmissions will be captured in the application and the EMR. For patients readmitted to Michigan Medicine, readmission parameters (reason for readmission, length of stay, interventions, ICU admission, etc.) will be captured and used to create a measure of readmission intensity. Descriptive statistics including (but not limited to) mean and standard deviation.

SECONDARY OUTCOMES:
Patient Experience Survey -- Application (all participants) | 42 days post hospital discharge
  Assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS®) GLOBAL 10 questionnaire.
Patient Experience Survey -- Application (first 20 participants) | 42 days post hospital discharge
  The first 20 participants will complete a qualtrix survey.
Readmission rate | 42 days post hospital discharge
  Readmissions will be captured in the application and the EMR. Descriptive statistics including (but not limited to) mean and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Montgomery, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No